CLINICAL TRIAL: NCT01426152
Title: Association Between Progesterone Levels on the Day of Ovulation Induction and IVF Outcome: Retrospective Study With 2500 Controlled Ovarian Stimulations Cycles
Brief Title: Progesterone on the Day of Ovulation Induction is Associated With Pregnancy Outcome
Acronym: ProgBBN
Status: Completed | Type: Observational
Sponsor: Bollmann Bruckner Noss (Other)
Responsible Party: Sponsor
Other Study IDs: Prog2006-2011; BBN (Other: Center for Reproductive Medicine)
Record Dates: First submitted 2011-08-28; First posted 2011-08-31 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Female Infertility
Keywords: IVF; progesterone; ovulation induction; pregnancy rates; Female Infertility Due to Nonimplantation
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Low level progesterone group (1): Progesterone < 1.50 ng/mL on day of ovulation induction
- Medium level progesterone group (2): Progesterone 1.51-1.99 ng/mL on the day of ovulation induction
- High level progesterone group (3): Progesterone > 1.99 ng/mL on the day of ovulation induction

SUMMARY:
Progesterone levels measured in blood/serum of patients on the day of ovulation induction following controlled ovarian stimulation for in vitro fertilization may be associated with pregnancy outcome. The hypothesis is that higher progesterone levels are associated with lower implantation rates due to changes in the endometrial receptivity.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ICSI following controlled ovarian stimulation
* progesterone measured on the day of ovulation induction
* informed consent

Exclusion Criteria:

* missing consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with infertility undergoing assisted reproduction techniques, i.e. in vitro fertilization.
Sampling Method: Probability Sample
Enrollment: 2555 (Actual)
Dates: Start 2006-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 13 weeks
  Patients will be followed up from embryotransfer until second trimester of pregnancy

SECONDARY OUTCOMES:
Delivery after 23.gestational weeks | 9 months
  Patients will be followed up from embryotransfer until delivery

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ochsenkuehn, MD, Principal Investigator — Center for Reproductive Medicine
Locations (1):
- Praxis Bollmann-Brückner-Noss, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Ochsenkuhn R, Arzberger A, von Schonfeldt V, Gallwas J, Rogenhofer N, Crispin A, Thaler CJ, Noss U. Subtle progesterone rise on the day of human chorionic gonadotropin administration is associated with lower live birth rates in women undergoing assisted reproductive technology: a retrospective study with 2,555 fresh embryo transfers. Fertil Steril. 2012 Aug;98(2):347-54. doi: 10.1016/j.fertnstert.2012.04.041. Epub 2012 May 24. PMID 22633265